CLINICAL TRIAL: NCT07250048
Title: A Randomised, Single-blind, Placebo-controlled Trial to Investigate Safety, Tolerability, and Pharmacokinetics of Single Rising Doses of BI 3009947 Administered Orally to Healthy Male Trial Participants, and a Randomised, Open-label, Single-dose, Three-way Cross-over Relative Bioavailability Comparison of Two Different Formulations for Oral Administration of BI 3009947 and the Effect of Food on One of These Formulations in Healthy Male Trial Participants
Brief Title: A Study in Healthy Men to Find Out How Different Doses of BI 3009947 Are Tolerated and How Different Formulations or Food Influence How BI 3009947 is Taken up Into the Blood
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1533-0001; 2025-521095-66-00 (Registry Identifier: CTIS); U1111-1318-3257 (Registry Identifier: WHO - International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: SRD part: placebo-controlled BA part: three-way crossover trial with 3 treatment periods to compare the relative bioavailability of reference treatment R and test treatments T1 and T2
Masking Description: SRD part: participants masked, single blind BA part: no masking, open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- SRD part: BI 3009947 Dose group 1 (Experimental)
  Interventions: Drug: BI 3009947 (Formulation A)
- SRD part: BI 3009947 Dose group 2 (Experimental)
  Interventions: Drug: BI 3009947 (Formulation A)
- SRD part: BI 3009947 Dose group 3 (Experimental)
  Interventions: Drug: BI 3009947 (Formulation A)
- SRD part: BI 3009947 Dose group 3fed (Experimental)
  Interventions: Drug: BI 3009947 (Formulation A)
- SRD part: BI 3009947 Dose group 4 (Experimental)
  Interventions: Drug: BI 3009947 (Formulation A)
- SRD part: BI 3009947 Dose group 4fed (Experimental)
  Interventions: Drug: BI 3009947 (Formulation A)
- SRD part: BI 3009947 Dose group 5 (Experimental)
  Interventions: Drug: BI 3009947 (Formulation A)
- SRD part: BI 3009947 Dose group 5fed (Placebo Comparator)
  Interventions: Drug: BI 3009947 (Formulation A)
- SRD part: BI 3009947 Dose group 6 (Experimental)
  Interventions: Drug: BI 3009947 (Formulation A)
- SRD part: BI 3009947 Dose group 6fed (Experimental)
  Interventions: Drug: BI 3009947 (Formulation A)
- SRD part: BI 3009947 Dose group 7 (Experimental)
  Interventions: Drug: BI 3009947 (Formulation A)
- SRD part: BI 3009947 Dose group 7fed (Experimental)
  Interventions: Drug: BI 3009947 (Formulation A)
- SRD part: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- BA part: Treatment sequence R-T1-T2 (Experimental): Reference treatment R and test treatments T1 and T2.
  Interventions: Drug: BI 3009947 (Formulation A); Drug: BI 3009947 (Formulation B)
- BA part: Treatment sequence T1-R-T2 (Experimental): Reference treatment R and test treatments T1 and T2.
  Interventions: Drug: BI 3009947 (Formulation A); Drug: BI 3009947 (Formulation B)
- BA part: Treatment sequence T2-R-T1 (Experimental): Reference treatment R and test treatments T1 and T2.
  Interventions: Drug: BI 3009947 (Formulation A); Drug: BI 3009947 (Formulation B)

INTERVENTIONS:
Drug: BI 3009947 (Formulation A) — BI 3009947 (Formulation A)
  Arms: BA part: Treatment sequence R-T1-T2; BA part: Treatment sequence T1-R-T2; BA part: Treatment sequence T2-R-T1; SRD part: BI 3009947 Dose group 1; SRD part: BI 3009947 Dose group 2; SRD part: BI 3009947 Dose group 3; SRD part: BI 3009947 Dose group 3fed; SRD part: BI 3009947 Dose group 4; SRD part: BI 3009947 Dose group 4fed; SRD part: BI 3009947 Dose group 5; SRD part: BI 3009947 Dose group 5fed; SRD part: BI 3009947 Dose group 6; SRD part: BI 3009947 Dose group 6fed; SRD part: BI 3009947 Dose group 7; SRD part: BI 3009947 Dose group 7fed
Drug: BI 3009947 (Formulation B) — BI 3009947 (Formulation B)
  Arms: BA part: Treatment sequence R-T1-T2; BA part: Treatment sequence T1-R-T2; BA part: Treatment sequence T2-R-T1
Drug: Placebo — Placebo matching BI 3009947 (Formulation A)
  Arms: SRD part: Placebo

SUMMARY:
Single-rising dose (SRD) part:

The main objectives of the SRD part of this trial are to investigate safety, tolerability, and pharmacokinetics (PK) of BI 3009947 in healthy participants following oral administration of single rising doses.

Bioavailability (BA) part:

The main objective of the BA part is to investigate the relative bioavailability of two different BI 3009947 formulations (Formulation A and B) and to assess the influence of food on the relative bioavailability of Formulation A or B.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male trial participant according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
2. Age of 18 to 45 years (inclusive)
3. Body mass index (BMI) of 18.5 to 29.9 kg/m^2 (inclusive)
4. Signed and dated written informed consent in accordance with international council for harmonisation-good clinical practice (ICH-GCP) and local legislation prior to admission to the trial

Exclusion Criteria:

1. Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
2. Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm
3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
4. Any evidence of a concomitant disease. This does not include acceptable concomitant conditions that were not assessed as clinically relevant by the investigator (e.g. possible cases of myopia, hyperopia, astigmatism, non-active pollinosis, or mild acne of the skin)
5. Further exclusion criteria apply.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-11-21 (Actual); Primary Completion 2026-05-13 (Estimated); Study Completion 2026-05-18 (Estimated)

PRIMARY OUTCOMES:
SRD part: Occurrence of any treatment-emergent adverse event assessed as drug-related by the investigator | up to Day 14
  This is expressed as the percentage of subjects treated with investigational drug who experience such an event.
BA part: AUC0-24 (area under the concentration-time curve of BI 3009947 in plasma over the dosing interval 0 to 24 hours) | up to Day 3
BA part: AUC0-24 (area under the concentration-time curve of the metabolite BI 3037996 in plasma over the dosing interval 0 to 24 hours) | up to Day 3
BA part: Cmax (maximum measured concentration of BI 3009947 in plasma) | up to Day 3
BA part: Cmax (maximum measured concentration of the metabolite BI 3037996 in plasma) | up to Day 3

SECONDARY OUTCOMES:
SRD part: AUC0-24 (area under the concentration-time curve of BI 3009947 in plasma over the dosing interval 0 to 24 hours) | up to Day 3
SRD part: AUC0-24 (area under the concentration-time curve of the metabolite BI 3037996 in plasma over the dosing interval 0 to 24 hours) | up to Day 3
SRD part: Cmax (maximum measured concentration of BI 3009947 in plasma) | up to Day 3
SRD part: Cmax (maximum measured concentration of the metabolite BI 3037996 in plasma) | up to Day 3
BA part: AUC0-∞ (area under the concentration-time curve of BI 3009947 in plasma over the time interval from 0 extrapolated to infinity) | up to Day 3
BA part: AUC0-∞ (area under the concentration-time curve of the metabolite BI 3037996 in plasma over the time interval from 0 extrapolated to infinity) | up to Day 3

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com